CLINICAL TRIAL: NCT01522976
Title: A Randomized Phase II/III Study of Azacitidine in Combination With Lenalidomide (NSC-703813) vs. Azacitidine Alone vs. Azacitidine in Combination With Vorinostat (NSC-701852) for Higher-Risk Myelodysplastic Syndromes (MDS) and Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Azacitidine With or Without Lenalidomide or Vorinostat in Treating Patients With Higher-Risk Myelodysplastic Syndromes or Chronic Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00242; NCI-2012-00242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000723909; SWOG-S1117; S1117 (Other: SWOG); S1117 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myelomonocytic Leukemia; Chronic Myelomonocytic Leukemia-1; Chronic Myelomonocytic Leukemia-2; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome/Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; GATA2 Deficiency | interventions — Azacitidine; Lenalidomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (azacitidine and lenalidomide) (Experimental): Patients receive azacitidine SC or IV on days 1-7 or days 1-5 and 8-9, and lenalidomide PO QD on days 1-21. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm II (azacitidine) (Experimental): Patients receive azacitidine as in Arm I. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis
- Arm III (azacitidine and vorinostat) (Experimental): Patients receive azacitidine as in Arm I and vorinostat PO BID on days 3-9. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm I (azacitidine and lenalidomide)
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm III (azacitidine and vorinostat)

SUMMARY:
This randomized phase II/III trial studies how well azacitidine works with or without lenalidomide or vorinostat in treating patients with higher-risk myelodysplastic syndromes or chronic myelomonocytic leukemia. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, stopping them from dividing, or by stopping them from spreading. Lenalidomide may stop the growth of cancer cells by stopping blood flow to the cancer. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether azacitidine is more effective with or without lenalidomide or vorinostat in treating myelodysplastic syndromes or chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To select based on response rate (complete remission, partial remission, or hematologic improvement) either the combination of lenalidomide and azacitidine or the combination of vorinostat and azacitidine for further testing against single-agent azacitidine among patients with higher-risk myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML). (Phase II) II. To compare overall survival between the combination arm selected in the Phase II portion of the trial to single-agent azacitidine among patients with higher-risk myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML). (Phase III)

SECONDARY OBJECTIVES:

I. To estimate relapse-free survival, overall survival and cytogenetic response rate of patients treated on each regimen.

II. To estimate the frequency and severity of toxicities of the three regimens in this patient population.

III. To investigate in a preliminary manner the frequency of subgroups from prestudy cytogenetic studies and correlate these subgroups with clinical outcomes in this patient population.

IV. To collect specimens for banking for use in future research studies.

TERTIARY OBJECTIVES:

I. To evaluate the prevalence of a pre-specified list of molecular lesions (48 total lesions).

II. To assess associations of these lesions with outcomes (response, event-free survival, relapse-free survival, and overall survival).

III. To develop a deoxyribonucleic acid (DNA) methylation biomarker predictive of response to DMTi treatment in MDS.

IV. To harness gene expression profiles as clinical biomarkers of primary resistance to DMTi in MDS.

OUTLINE: Patients are randomized to 1 of 3 treatment arms. In Phase III, patients are randomized to 1 of 2 treatment arms (the combination arm selected in Phase II or the single-agent azacitidine arm).

ARM I: Patients receive azacitidine subcutaneously (SC) or intravenously (IV) on days 1-7 or days 1-5 and 8-9, and lenalidomide orally (PO) once daily (QD) on days 1-21.

ARM II: Patients receive azacitidine as in Arm I.

ARM III: Patients receive azacitidine as in Arm I and vorinostat PO twice daily (BID) on days 3-9.

In all arms, treatment repeats every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have morphologically confirmed diagnosis of myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) based on one of the following:

  * French-American-British (FAB) classifications:

    * Refractory anemia with excess blasts (RAEB - defined as having 5-20% myeloblasts in the bone marrow)
    * Chronic myelomonocytic leukemia (CMML) with 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood
  * World Health Organization (WHO) classifications:

    * Refractory anemia with excess blasts-1 (RAEB-1 - defined as having 5-9% myeloblasts in the bone marrow)
    * Refractory anemia with excess blasts-2 (RAEB-2 - defined as having 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood)
    * Chronic myelomonocytic leukemia-1 (CMML-1 - defined as having < 10% myeloblasts in the bone marrow and/or < 5% blasts in the blood)
    * Chronic myelomonocytic leukemia-2 (CMML-2 - defined as having 10-19% myeloblasts in the bone marrow and/or 5-19% blasts in the blood) OR
  * International prognostic score (IPSS) of intermediate 2 (1.5-2.0 points) or high (>= 2.5 points); a score of intermediate 1 (0.5-1.0 points) is only allowable in the setting of >= 5% myeloblasts
  * NOTE: Patients with acute myeloid leukemia (AML) are not eligible
  * Procedures to obtain specimens for establishing baseline disease must be done within 30 days prior to registration
* Patients must not have received lenalidomide, azacitidine, vorinostat, or decitabine as treatment previously; any hematopoietic growth factors must be stopped for at least 14 days prior to registration; patients may have received low-dose cytarabine for MDS treatment previously, but they must have discontinued its use for at least 28 days prior to registration; patients may have received prior hydroxyurea per CMML treatment previously, but they must have discontinued its use for at least 7 days prior to registration; these patients will not be eligible if white blood cell (WBC) > 30,000/mm^3
* Patients must not have received radiation therapy, chemotherapy, or cytotoxic therapy to treat conditions other than MDS within 12 months prior to registration
* Patients must not have undergone prior allogeneic stem cell or bone marrow transplantation at any time; patients that have undergone an autologous stem cell transplant are eligible
* Patients must not have used or be using histone deacetylase (HDAC) inhibitor agents for anticancer treatment
* Patients may not have received agents such as valproic acid for epilepsy within 30 days prior to registration
* Patients must have Zubrod performance status of 0-2
* Patients must not have any pre-existing neurotoxicity/neuropathy of >= grade 2 according to the National Cancer Institute (NCI) Common Toxicity Criteria version 4.0, or prior >= grade 3 allergic reaction/hypersensitivity or rash to thalidomide, that has not resolved to < grade 2
* Patients must not have any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent
* Patients must not have history of thromboembolic event or other condition requiring current use of anticoagulation with Coumadin (warfarin) or low molecular-weight heparin
* Patients must not have known or suspected hypersensitivity to mannitol
* Patients must receive a 12-lead electrocardiogram (EKG), chest x-ray or computed tomography (CT) scan, serum creatinine, complete metabolic panel including serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT), electrolytes, and bilirubin testing within 28 days prior to registration in order to establish baseline measurements; questions regarding patient safety in regards to results of these tests should be directed to the study chair
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to registration; FCBP must agree to have a second pregnancy test within 24 hours prior to starting cycle 1 if randomized to receive lenalidomide

  * Further, patients commit to the following if they are randomized to receive lenalidomide: FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
  * NOTE: Patients not randomized to receive lenalidomide will not be required to undergo serial pregnancy testing or lenalidomide counseling after registration
* No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for three years
* Cytogenetics requirements:

  * Southwestern Oncology Group (SWOG) (and other sites not affiliated with Alliance or Eastern Cooperative Oncology Group [ECOG]-American College of Radiology Imaging Network [ACRIN]): Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 30 days prior to registration to S1117; specimens must be submitted to the site's preferred Clinical Laboratory Improvement Amendments (CLIA)-approved cytogenetics laboratory; reports of the results must be submitted as described; note that cytogenetics are required at other timepoints; NOTE: National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) sites may submit specimens to College of American Pathologists (CAP) or Ontario Laboratory Accreditation (OLA)-approved laboratories providing the lab is licensed to perform fluorescent in situ hybridization (FISH) analysis
  * Alliance: Alliance patients must enroll on Cancer and Leukemia Group B (CALGB) 8461, the cytogenetics protocol; CALGB 8461 provides sample procurement and submission instructions to Alliance-approved institutional cytogeneticists; note that cytogenetics are required at other timepoints
  * ECOG-ACRIN: Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 30 days prior to registration to S1117; specimens must be submitted to the site's preferred CLIA-approved cytogenetics laboratory; karyotypes and reports must be submitted for review to the Mayo Clinic Cytogenetics Laboratory in Rochester; note that cytogenetics testing is required at other timepoints
* Banking requirements:

  * SWOG, Alliance and ECOG-ACRIN (and other sites not affiliated with NCIC CTG): Patients must be offered participation in specimen banking; with patient consent, specimens must be submitted as outlined
  * Alliance: (Temporarily Closed 2/28/14): As of February 28, 2014, CALGB 9665 has been temporarily closed, so Alliance patients under consideration for S1117 are NOT to be registered to CALGB 9665 and no specimens for patients enrolled after February 28, 2014 are to be submitted via this ancillary study; these patients should submit specimens per SWOG instructions; patients already enrolled on CALGB 9665 should continue to submit specimens per instructions in CALGB 9665
  * NCIC CTG: NCIC CTG patients must be offered participation in specimen submission and banking; with patient consent, specimens must be submitted as outlined
* All patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael A Sekeres, Principal Investigator — SWOG Cancer Research Network
Locations (294):
- United States (280):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center -Washington DC, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Sovah Health Martinsville, Martinsville, Virginia
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (14):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Clinical Research Unit at Vancouver Coastal Health Authority, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Statler A, Othus M, Erba HP, Chauncey TR, Radich JP, Coutre S, Advani A, Nand S, Ravandi F, Mukherjee S, Sekeres MA. Comparable outcomes of patients eligible vs ineligible for SWOG leukemia studies. Blood. 2018 Jun 21;131(25):2782-2788. doi: 10.1182/blood-2018-01-826693. Epub 2018 Apr 4. PMID 29618479

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Azacitidine/Lenalidomide: Patients receive azacitidine SC or IV on days 1-7 or days 1-5 and 8-9, and lenalidomide PO QD on days 1-21. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given SC or IV
  Lenalidomide: Given PO
- Arm 2: Azacitidine: Patients receive azacitidine as in Arm 1. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given SC or IV
- Arm 3: Azacitidine/Vorinostat: Patients receive azacitidine as in Arm 1 and vorinostat PO BID on days 3-9. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given SC or IV
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Started | 97 | 92 | 93
Completed | 0 | 0 | 0
Not Completed | 97 | 92 | 93
Not completed — Ineligible | 4 | 0 | 1
Not completed — Death | 7 | 6 | 2
Not completed — Still on treatment | 9 | 9 | 6
Not completed — Disease progression | 28 | 30 | 25
Not completed — Adverse Event | 17 | 7 | 18
Not completed — Refusal unrelated to adverse event | 10 | 13 | 14
Not completed — Not protocol specified | 22 | 27 | 27

BASELINE CHARACTERISTICS:
Population: Analysis includes eligible patients only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat | Total
Number analyzed (Participants) | 93 | 92 | 92 | 277
Age, Continuous [Median (Full Range); unit: years] | 70.81 [51.29 to 86.68] | 69.67 [42.69 to 88.96] | 70.36 [28.69 to 93.01] | 70.18 [28.69 to 93.01]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 22 | 85
  Male | 61 | 61 | 70 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 4 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 3 | 4 | 9
  White | 86 | 80 | 83 | 249
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Phase II)
Description: A response is any of complete hematological remission, partial remission, or hematologic improvement.
Time Frame: Up to 5 years
Population: Analysis includes eligible patients only.
Measure: Number (95% Confidence Interval); unit: percentage of patients having a response
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 93 | 92 | 92
percentage of patients having a response | 49 [39 to 60] | 38 [28 to 49] | 27 [18 to 37]

2. Primary Outcome: Overall Survival (Phase III)
Description: OS is calculated for all patients from the date of initial registration to date of death due to any cause. The follow-up for patients last known to be alive is censored at the date of last contact. Stratified Cox regression models will be used to compare OS of the combination arm selected in the Phase II portion of the trial to OS of the single-agent azacitidine arm.
Time Frame: Up to 5 years
Population: This trial did not proceed to the Phase III portion. Therefore, no patients were analyzed for this outcome measure.
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Relapse-free Survival
Description: RFS is calculated for patients who have achieved a response. RFS will be measured from the date of response to the date of first documentation of relapse from response (as defined in the primary objective), or death due to any cause. The follow-up for patients last known to be alive and without report of relapse is censored at the date of last contact. RFS will be estimated for each of the three arms using the Kaplan-Meier method.
Time Frame: Up to 5 years
Population: Analysis includes eligible patients who had a response.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 46 | 35 | 25
Days | 435 [237 to 546] | 311 [182 to 640] | 455 [197 to NA] — The upper limit of the confidence interval cannot be estimated.

4. Secondary Outcome: Overall Survival
Description: OS is calculated for all patients from the date of initial registration to date of death due to any cause. The follow- up for patients last known to be alive is censored at the date of last contact. OS will be estimated for each of the three arms using the Kaplan-Meier method.
Time Frame: Up to 5 years
Population: Analysis includes eligible patients only.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 93 | 92 | 92
Days | 588 [426 to 737] | 449 [356 to 603] | 527 [392 to 852]

5. Secondary Outcome: Pre-study Cytogenetic Abnormalities
Description: Cytogenetic risk group is used to identify cytogenetic abnormalities.
Time Frame: Up to 5 years
Population: Analysis includes eligible patients only.
Measure: Number; unit: participants
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 93 | 92 | 92
participants
  Good/very good | 35 | 29 | 34
  Intermediate | 13 | 16 | 18
  Poor | 8 | 10 | 8
  Very poor | 23 | 23 | 19
  Missing | 14 | 14 | 13

6. Secondary Outcome: Toxicity Rate
Description: Adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Analysis includes only eligible patients who also received treatment.
Measure: Number; unit: Participants
Groups:
- Arm 1: Azacitidine/Lenalidomide: Patients receive azacitidine SC or IV on days 1-7 or days 1-5 and 8-9, and lenalidomide PO QD on days 1-21. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Azacitidine: Given SC or IV
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Number analyzed (Participants) | 89 | 91 | 91
Participants
  Abdominal infection | 1 | 0 | 0
  Abdominal pain | 1 | 0 | 3
  Acute kidney injury | 0 | 0 | 1
  Adult respiratory distress syndrome | 1 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 5
  Anemia | 48 | 37 | 44
  Anorectal infection | 0 | 0 | 1
  Anorexia | 4 | 0 | 3
  Apnea | 0 | 0 | 1
  Ascites | 1 | 0 | 1
  Aspartate aminotransferase increased | 0 | 0 | 3
  Ataxia | 0 | 0 | 1
  Back pain | 1 | 0 | 0
  Blood and lymphatic system disorders - Other | 0 | 2 | 1
  Blood bilirubin increased | 0 | 0 | 3
  Bronchial infection | 0 | 0 | 1
  CD4 lymphocytes decreased | 1 | 0 | 0
  Cardiac arrest | 1 | 0 | 0
  Catheter related infection | 1 | 2 | 1
  Cecal infection | 0 | 0 | 1
  Cholecystitis | 0 | 0 | 1
  Colitis | 0 | 0 | 1
  Confusion | 0 | 0 | 1
  Constipation | 2 | 1 | 1
  Creatinine increased | 2 | 0 | 0
  Dehydration | 5 | 1 | 3
  Delirium | 0 | 0 | 1
  Diarrhea | 5 | 0 | 3
  Dizziness | 1 | 0 | 0
  Dyspnea | 4 | 2 | 3
  Epistaxis | 0 | 0 | 1
  Esophageal pain | 0 | 0 | 1
  Esophagitis | 1 | 0 | 0
  Fall | 0 | 0 | 1
  Fatigue | 9 | 6 | 14
  Febrile neutropenia | 16 | 11 | 13
  Fever | 0 | 0 | 2
  Flushing | 0 | 0 | 1
  Gastric hemorrhage | 0 | 0 | 1
  Gastrointestinal pain | 1 | 0 | 1
  General disorders and admin site conditions-Other | 1 | 0 | 0
  Generalized muscle weakness | 3 | 1 | 3
  Hallucinations | 0 | 0 | 1
  Headache | 0 | 0 | 1
  Heart failure | 0 | 0 | 1
  Hematoma | 0 | 0 | 1
  Hematuria | 1 | 0 | 2
  Hyperglycemia | 1 | 1 | 2
  Hypernatremia | 0 | 1 | 0
  Hypertension | 1 | 0 | 2
  Hyperuricemia | 0 | 0 | 1
  Hypoalbuminemia | 3 | 0 | 0
  Hypokalemia | 4 | 0 | 1
  Hypomagnesemia | 1 | 0 | 0
  Hyponatremia | 5 | 1 | 4
  Hypophosphatemia | 1 | 0 | 2
  Hypotension | 4 | 0 | 3
  Hypoxia | 0 | 0 | 1
  Infections and infestations - Other, specify | 4 | 2 | 5
  Intracranial hemorrhage | 1 | 0 | 0
  Investigations - Other, specify | 1 | 0 | 0
  Leukocytosis | 0 | 1 | 0
  Lower gastrointestinal hemorrhage | 0 | 0 | 2
  Lung infection | 4 | 1 | 2
  Lymphocyte count decreased | 14 | 9 | 3
  Lymphocyte count increased | 0 | 1 | 1
  Mucosal infection | 0 | 0 | 1
  Mucositis oral | 1 | 0 | 0
  Nausea | 1 | 2 | 2
  Neutrophil count decreased | 69 | 48 | 63
  Pain | 1 | 0 | 0
  Papulopustular rash | 1 | 0 | 0
  Pericardial effusion | 1 | 0 | 0
  Platelet count decreased | 61 | 46 | 64
  Pneumonitis | 0 | 0 | 1
  Pruritus | 1 | 0 | 0
  Pulmonary edema | 0 | 0 | 1
  Purpura | 1 | 0 | 0
  Rash maculo-papular | 13 | 3 | 1
  Renal and urinary disorders - Other, specify | 0 | 0 | 1
  Respiratory failure | 0 | 0 | 1
  Sepsis | 4 | 2 | 3
  Sinus bradycardia | 1 | 0 | 0
  Skin infection | 3 | 1 | 2
  Soft tissue infection | 1 | 1 | 0
  Sudden death NOS | 0 | 1 | 0
  Syncope | 2 | 0 | 4
  Thromboembolic event | 1 | 0 | 1
  Tooth infection | 0 | 0 | 1
  Upper gastrointestinal hemorrhage | 0 | 0 | 1
  Upper respiratory infection | 0 | 1 | 0
  Urinary tract infection | 1 | 1 | 1
  Vascular disorders - Other, specify | 0 | 0 | 1
  Vomiting | 1 | 1 | 1
  Weight loss | 1 | 0 | 0
  White blood cell decreased | 48 | 34 | 44

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Analysis includes only eligible patients who also received treatment. Adverse events that are possibly, probably or definitely related to study drug are reported.
Arm/Group | Arm 1: Azacitidine/Lenalidomide | Arm 2: Azacitidine | Arm 3: Azacitidine/Vorinostat
Serious Adverse Events (participants affected / at risk) | 37/89 | 8/91 | 47/91
Other Adverse Events (participants affected / at risk) | 88/89 | 89/91 | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Azacitidine/Lenalidomide (N=89) | Arm 2: Azacitidine (N=91) | Arm 3: Azacitidine/Vorinostat (N=91)
Anemia (Blood and lymphatic system disorders) | 6 | 0 | 6
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 2
Heart failure (Cardiac disorders) | 1 | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 4
Fever (General disorders) | 1 | 0 | 6
Infusion related reaction (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Sudden death NOS (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 2 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 1
Infections and infestations-Other (Infections and infestations) | 4 | 0 | 8
Lip infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 5 | 0 | 4
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 2 | 4
Skin infection (Infections and infestations) | 2 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 2
Investigations-Other (Investigations) | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 4
Platelet count decreased (Investigations) | 7 | 0 | 8
White blood cell decreased (Investigations) | 3 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 2 | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 4
Confusion (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 3 | 0 | 3
Thromboembolic event (Vascular disorders) | 1 | 0 | 1
Vascular disorders-Other (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Azacitidine/Lenalidomide (N=89) | Arm 2: Azacitidine (N=91) | Arm 3: Azacitidine/Vorinostat (N=91)
Anemia (Blood and lymphatic system disorders) | 76 | 71 | 72
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 14 | 13
Chest pain - cardiac (Cardiac disorders) | 3 | 2 | 6
Sinus tachycardia (Cardiac disorders) | 3 | 4 | 9
Abdominal pain (Gastrointestinal disorders) | 8 | 14 | 21
Constipation (Gastrointestinal disorders) | 49 | 54 | 44
Diarrhea (Gastrointestinal disorders) | 42 | 23 | 53
Dry mouth (Gastrointestinal disorders) | 10 | 9 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 13 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 6
Hemorrhoids (Gastrointestinal disorders) | 5 | 2 | 4
Mucositis oral (Gastrointestinal disorders) | 15 | 7 | 10
Nausea (Gastrointestinal disorders) | 38 | 42 | 61
Oral pain (Gastrointestinal disorders) | 5 | 2 | 4
Vomiting (Gastrointestinal disorders) | 18 | 18 | 36
Chills (General disorders) | 19 | 11 | 10
Edema limbs (General disorders) | 24 | 22 | 28
Fatigue (General disorders) | 74 | 69 | 74
Fever (General disorders) | 14 | 19 | 15
General disorders and admin site conditions - Other (General disorders) | 5 | 4 | 5
Injection site reaction (General disorders) | 22 | 19 | 18
Non-cardiac chest pain (General disorders) | 2 | 3 | 5
Pain (General disorders) | 14 | 10 | 10
Infections and infestations-Other (Infections and infestations) | 9 | 10 | 8
Lung infection (Infections and infestations) | 2 | 6 | 5
Skin infection (Infections and infestations) | 9 | 13 | 9
Upper respiratory infection (Infections and infestations) | 5 | 6 | 4
Urinary tract infection (Infections and infestations) | 8 | 2 | 3
Bruising (Injury, poisoning and procedural complications) | 25 | 24 | 18
Fall (Injury, poisoning and procedural complications) | 0 | 6 | 7
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 2 | 5 | 0
Alanine aminotransferase increased (Investigations) | 18 | 16 | 17
Alkaline phosphatase increased (Investigations) | 17 | 16 | 13
Aspartate aminotransferase increased (Investigations) | 18 | 23 | 17
Blood bilirubin increased (Investigations) | 14 | 13 | 24
Creatinine increased (Investigations) | 21 | 26 | 25
INR increased (Investigations) | 4 | 5 | 3
Lymphocyte count decreased (Investigations) | 32 | 16 | 19
Neutrophil count decreased (Investigations) | 77 | 58 | 73
Platelet count decreased (Investigations) | 78 | 68 | 69
Weight loss (Investigations) | 22 | 15 | 19
White blood cell decreased (Investigations) | 66 | 52 | 60
Anorexia (Metabolism and nutrition disorders) | 39 | 31 | 45
Dehydration (Metabolism and nutrition disorders) | 9 | 10 | 17
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 6 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 33 | 27 | 32
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 6 | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 7 | 5
Hypernatremia (Metabolism and nutrition disorders) | 5 | 3 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 5 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 29 | 21 | 32
Hypocalcemia (Metabolism and nutrition disorders) | 30 | 16 | 25
Hypokalemia (Metabolism and nutrition disorders) | 40 | 15 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 10 | 9
Hyponatremia (Metabolism and nutrition disorders) | 23 | 22 | 34
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 11 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 18 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 22 | 15 | 23
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 12 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 16 | 12
Dizziness (Nervous system disorders) | 19 | 22 | 28
Dysgeusia (Nervous system disorders) | 11 | 11 | 16
Headache (Nervous system disorders) | 12 | 14 | 16
Paresthesia (Nervous system disorders) | 5 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 10 | 8
Tremor (Nervous system disorders) | 5 | 3 | 2
Anxiety (Psychiatric disorders) | 15 | 13 | 6
Confusion (Psychiatric disorders) | 3 | 5 | 4
Depression (Psychiatric disorders) | 9 | 9 | 12
Insomnia (Psychiatric disorders) | 18 | 15 | 14
Chronic kidney disease (Renal and urinary disorders) | 1 | 3 | 7
Proteinuria (Renal and urinary disorders) | 4 | 7 | 1
Urinary frequency (Renal and urinary disorders) | 5 | 2 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 26 | 28
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 41 | 36 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 13 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 15 | 7
Purpura (Skin and subcutaneous tissue disorders) | 6 | 5 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 46 | 20 | 16
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 14 | 15 | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 | 1 | 6
Hematoma (Vascular disorders) | 5 | 4 | 5
Hot flashes (Vascular disorders) | 9 | 4 | 5
Hypertension (Vascular disorders) | 10 | 11 | 11
Hypotension (Vascular disorders) | 13 | 5 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less